CLINICAL TRIAL: NCT07166952
Title: Peripheral Nerve Stimulation With the SPRINT® System in Chronic Posterior Sacroiliac Joint Complex Pain
Brief Title: Peripheral Nerve Stimulation With the SPRINT® System in Chronic PSIJC Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: SPR Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Ameet Nagpal, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00140724
Record Dates: First submitted 2025-09-09; First posted 2025-09-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SPRINT PNS System for chronic lower back pain (Experimental): This study will observe changes in pain intensity and functional status using the Numeric Rating Scale (NRS) and Oswestry Disability Index (ODI) over a 3-month follow-up period.
  Interventions: Device: SPRINT PNS System

INTERVENTIONS:
Device: SPRINT PNS System — This study will evaluate patient-reported outcomes, including pain and function, following standard clinical use of the SPRINT PNS System for posterior sacroiliac joint complex (PSIJC) pain.

SUMMARY:
Chronic lower back pain is a significant cause of disability, affecting 21-68% of people 60 years of age and older (source). Of these cases, 15-30% are attributed to posterior sacroiliac joint complex (PSIJC) pain (source), making it a target for treatment. Peripheral Nerve Stimulation (PNS) is a procedure that involves the placement of a lead under the skin with local anesthetic and electrically stimulating designated spinal nerves that deliver pain signals to the brain. It has emerged as a promising alternative to drug, injection, and radioablative therapies. Its use has been supported by previous studies of subjects who received permanent neurostimulation and experienced benefits such as decreased sensation of pain and perceived level of disability. SPRINT is a minimally invasive PNS system of interest due to its ability to provide long-term pain relief after temporary administration of PNS. The aim of this study is to understand whether the FDA-cleared SPRINT PNS system is safe and effective for the treatment of chronic PSIJC pain. This prospective clinical study will assess 10 subjects that meet the inclusion and exclusion criteria across 5 separate time points- 1.) Screening; 2.) Procedure within 3 months of screening; 3.) 12-day post-procedure follow-up; 4.) 3-month post-procedure follow-up; 5.) 3-Month post lead removal follow-up. The subjects will be required to complete physical examinations, and VAS and ODI questionnaires at timepoints 3, 4, and 5.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a leading cause of disability in the United States, with a recent review finding a prevalence between 21-68% of all people aged 60 or older. Posterior sacroiliac joint complex (PSIJC) pain affects a large percentage of these patients, with a prevalence of 15-30% of all CLBP cases. The etiology of sacroiliac dysfunction is complex and often includes multiple factors. Patients may experience pain from inflammation of the SI joint itself, or dysfunction of the supporting tendons and ligaments may produce pain by affecting the ability of the joint to effectively transfer loads. The verbiage used for this clinical syndrome has been altered to PSIJC to include the posterior connective tissues as a consideration in the diagnosis and treatment. The cause of pain may be from the joint itself, associated tendons, muscles, or a combination of sources. The innervation of the sacroiliac complex is extensive, but a large component of the posterior complex innervation is from the lateral branches of the sacral dorsal rami. The gold standard for diagnosis has been analgesic response to SIJ injection with local anesthetic. Therapeutic injections of the joint are utilized, but reimbursement from payors has been restricted due to the small sample sizes and limited difference in pain medication use and functional improvement. Since the restrictions on therapeutic injections, radiofrequency ablation has become a mainstay interventional modality.

Sacral lateral branch radiofrequency ablation (SLBRFA) has been used to treat PSIJC pain for many years, with multiple studies finding a majority of subjects receiving ≥50% relief at 1, 3, 6, and 12 months. One study examining the effectiveness of endoscopic radiofrequency ablation of PSIJC for CLBP found a 61% reduction in Visual Analog Scale (VAS) score and 50% reduction in Oswestry Disability Index (ODI) at 24 months following the procedure. Despite the evidence for utilizing SLBRFA to treat PSIJC pain, on March 19, 2023, the Centers for Medicare & Medicaid Services (CMS) joined private payors in deeming SLBRFA as "not reasonable and necessary," all but eliminating access to this treatment for most Americans. The rationale for no longer covering SLBRFA includes a lack of high-quality evidence for SLBRFA over placebo for PSIJC pain, as studies conducted have been hindered by small sample sizes and variability in patient selection and procedure technique. They also noted remaining concerns over the safety profile of this procedure and the lack of clear diagnostic criteria for determining patients that will benefit from SLBRFA. Unfortunately, the denial of access to SLBRFA has left a gap regarding interventional solutions in the treatment of PSIJC pain. Symptoms are often refractory to medical and physiotherapies and the evidence for these modalities is limited by small sample sizes and a limited number of studies. Recent evidence for spinal cord stimulation for non-surgical low back pain made headlines, however PSIJC pain has never specifically been examined. There is great concern among physicians treating this disease that the lack of less invasive treatment options will result in more unnecessary or ineffective SIJ fusions.14 SIJ fusion technology has been limited by conflicting data on efficacy, a complication rate of up to 16%, and the changing loads on the joint and surrounding structures after fusion. The lack of options also limits the ability to treat PSIJC pain in patients deemed to not be surgical candidates for SIJ fusion.

Unfortunately, interventional providers have little to offer those suffering from PSIJC pain in this new paradigm. An alternative is desperately needed for patients and providers prior to considering SIJ fusion. Previous studies have shown that peripheral nerve stimulation (PNS) can successfully treat multiple types of chronic pain. There is a nascent body of evidence for treating PSIJC pain with PNS, and this evidence has been promising. Notably, one trial of 16 patients by Guentchev et al. implanted a permanent neurostimulator targeting the S1-S3 lateral branches (Prime Advanced™ Medtronic, Dublin, Ireland) following a successful trial (>50% pain relief for up to 1 week). Results of this trial have demonstrated PNS to be effective as both a short term and long-term treatment of PSIJC pain, finding average ODI decreased to 23% from 58% at 1 year and average VAS decreased to 1.6 and 2.0 (from 8.8 pre-implantation) at 1 and 3 years post-implantation, respectively. Similar effectiveness in treating intractable PSIJC pain with permanent neurostimulators has been shown in case reports. One case report involved a 41-year-old woman with PSIJC pain that was successfully treated (VAS decreased to 3 from 9) with permanent sacral nerve stimulation to the left first sacral foramen after she did not sustain lasting pain relief from intramuscular piriformis injection, SIJ intra-articular injection, and radiofrequency denervation. Another case report demonstrated permanent peripheral nerve field stimulation for SIJ pain was able to cut pain medication requirements by half while also providing >50% improvement in functional status in 2 patients who failed to receive >3 months of relief from injections or RFA. An interesting case report of a 74-year-old female with SIJ pain demonstrated the effectiveness of permanent neurostimulation via leads placed both epidurally and in the subcutaneous tissue overlying the bilateral SI joints. A three-day trial of epidural spinal cord stimulation yielded no improvement before a trial of subcutaneous field stimulation was performed with relief. She has received a 90% improvement in symptoms with a drop in her VAS from 10 to 1 and increased independence with her activities of daily living ongoing at 2 years. Lastly, there is also one randomized trial actively recruiting patients to SLB PNS versus best medical treatment in Germany.

While there is evidence permanent PNS can be effective and durable, temporary PNS for PSIJC pain has not been examined. Investigators have reason for optimism that the temporary SPRINT system may provide durable relief. The platform has demonstrated its utility and cost effectiveness in similar chronic pain syndromes. A trial performed by Gilmore et al. examined the long-term effectiveness after a 30-day implantation period of the percutaneous SPRINT PNS System (SPR Therapeutics) targeting the medial branches of the dorsal rami for the treatment of facetogenic CLBP. This trial demonstrated durable long-term relief at 12-months post-explanation, with 50% of participants having a clinically significant reduction (≥ 50%) in pain intensity and in disability as measured by the ODI. Given the recent changes in access to SLBRFA, combined with promising results of temporary PNS in treating chronic pain syndromes, further investigation into the effectiveness of temporary PNS for PSIJC pain is warranted. Investigators aim to examine the effectiveness of temporary sacral lateral branch PNS with the SPRINT® system as a minimally invasive long-term solution for the treatment PSIJC pain. To do this, investigators initially propose performing a ten patient prospective case series to prove the viability of the application and examine its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Sacroiliac pain as diagnosed above
* Subject greater than 18 years old
* Subject is severely debilitated by SIJ pain, with initial ODI score > 40%
* Subject received conservative treatment for at least three months including physiotherapy and pain medication
* Subject is able to understand and consent to the study and device management and participating in follow-up surveys
* Subject is scheduled for a commercial SPRINT case that has been authorized through their healthcare insurance

Exclusion Criteria:

* Pregnancy
* Subject is under the age of 18 years
* Acute traumatic injury of the sacral iliac joint
* Active inflammation or neoplastic infiltration of the SIJ
* Neoplastic diseases of the spine
* Spinal surgery within the last three months
* Sacroiliac joint steroid injection within the past 1 month or sacral lateral branch radiofrequency ablation within the past 6 months
* Contraindication for Neuromodulation Device (severe psychiatric disease, severe coagulation disorder, acute infection, active autoimmune disease with immunosuppression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-26 (Actual); Primary Completion 2027-10-26 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale at 60 days and 90 days post procedure (lead removal) | at 60 days (plus or minus 5 days) and 90 days (plus or minus 10 days)

SECONDARY OUTCOMES:
Measurement of the Oswestry Disability Index (ODI) at the 60 and 90 day post Lead removal | at 60 days (plus or minus 5 days) and 90 days (plus or minus 10 days) post Lead removal

CONTACTS AND LOCATIONS:
Overall Officials: Ameet Nagpal, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published in a scientific journal; individual data will not be shared.